CLINICAL TRIAL: NCT04218630
Title: Investigation Of Effectiveness Of Reformer Pilates In Individuals With Fibromyalgia: Randomized Controlled Trial
Brief Title: Pilates Exercises In Individuals With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berna Cagla Caglayan (Other)
Responsible Party: Sponsor-Investigator, Berna Cagla Caglayan, Principal Investigator, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787
Record Dates: First submitted 2019-12-31; First posted 2020-01-06 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
Keywords: Reformer pilates; Mat pilates; Fibromyalgia; Exercise
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled parallel group model. Participants were randomly divided into two groups as reformer pilates group and home mat pilates group.
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist performing evaluation was blind to the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer pilates group (Experimental): All participants were informed about the reformer machine and the treatment program by the physiotherapist in reformer pilates group. Reformer pilates exercises were applied in the form of general muscle strengthening and flexibility exercises under the supervision of physiotherapist. Exercises were performed in 2 times a week for 6 weeks. The duration of one session was 60 minutes.
  Interventions: Other: Reformer pilates exercises
- Home mat pilates group (Active Comparator): In home mat pilates group, clinical pilates exercises were applied as a home program. Brochures and exercise follow-up forms, which illustrated and written all the exercises in this program, which consisted of clinical pilates-based general muscle strength and flexibility exercises, were given to all participants in this group. Exercises were performed in 2 times a week for 6 weeks at home. Participants marked the follow-up form when they performed exercises. Attendance of participants to exercise was checked by phone calls.
  Interventions: Other: Home mat pilates exercises

INTERVENTIONS:
Other: Reformer pilates exercises — The program consisted of 10 minutes warm-up exercises, reformer pilates exercises for 40 minutes and 10 minutes cool-down exercises. The exercises were started with 6-8 repetitions, increased to 1-2 repetitions each week and applied to be 12-15 repetitions in the last week. Increasing the resistance of the springs and adding different positions were used for progression of exercises.
  Arms: Reformer pilates group
Other: Home mat pilates exercises — The program consisted of 10 minutes warm-up exercises, clinical pilates-based exercises on mat for 40 minutes and 10 minutes cool-down exercises. The exercises were started with 6-8 repetitions, increased to 1-2 repetitions each week, and applied to be 12-15 repetitions in the last week.
  Arms: Home mat pilates group

SUMMARY:
This study investigated the effects of reformer pilates exercises in Fibromyalgia, which is a chronic musculoskeletal disease characterized by widespread pain in the body, on number of painful regions, disease activity, lower extremity muscle strength, functional mobility, balance, kinesophobia, fatigue, sleep quality, biopsychosocial status and quality of life and compared effects of clinical pilates-based home pilates which is performed on a mat.

DETAILED DESCRIPTION:
In this study, effects of reformer pilates were evaluated by comparing with home mat pilates method. A total of 28 volunteer women who were diagnosed with FM according to the American College of Rheumatology (ACR) 2016 criteria were included in the study. Reformer pilates group had 14 participants, home mat pilates group had 14 participants.

All individuals were evaluated by same physiotherapist according to standardized test protocols and in the same conditions at baseline and at the end of 6th week. Number of painful regions with Pain Location Inventory (PLI), disease activity with Fibromyalgia Impact Questionnaire (FIQ), lower extremity muscle strength with Chair Test, functional mobility with The Timed Up and Go Test (TUG), balance with Single Leg Stance Test, kinesiophobia with Tampa Kinesiophobia Scale, fatigue with Fatigue Severity Scale, sleep quality with Pittsburgh Sleep Quality Index (PSQI), biopsychosocial status with Cognitive Exercise Therapy Approach- Biopsychosocial Questionnaire (BETY-BQ) and quality of life with Short Form-36 (SF-36) were evaluated.

Pilates exercises were performed by a certified and experienced physiotherapist in this field as two different methods (reformer group and home mat group) in 2 times a week for 6 weeks. Before starting treatment program, 5 key elements of clinical pilates exercises, which are breathing, focus, and placement of the rib cage, shoulder, head and neck, were taught to all patients. Participants were encouraged to focus and maintain these 5 key elements during all exercises.

Data were assessed using SPSS (Version 21.0). Continuous variables were stated as average, standard deviation and percentage. When parametric test assumptions were provided the Independent Samples Test was used, when parametric test assumptions were not provided Mann-Whitney U test was used to compare the differences between the independent groups. When parametric test assumptions were provided, the Paired Simple T Test was used, when parametric test assumptions were not provided, Wilcoxon signed-rank test was used to compare the differences between the dependent groups. P value <0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* having FM diagnosis according to ACR 2016 criteria
* aged 18-65
* being stable in drug use for at least 3 months or more
* being volunteer to participate in this study

Exclusion Criteria:

* doing exercise regularly for the last 3 months
* having orthopaedic and cardiopulmonary diseases which would prevent patients of doing exercise
* neurological disorders
* unstable endocrine system diseases
* malignancy, pregnancy
* severe psychological diseases
* having undergone any surgery in the last 6 months
* having communication problems.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 1 year
  It is a questionnaire consisting of 10 questions which assess physical health, work status, depression, anxiety, sleep, pain, fatigue, stiffness and well-being in order to evaluate health status and physical functionality of individuals with fibromyalgia.
Pain Location Inventory | 1 year
  Participants mark the areas in which feel pain in last seven days from the 28 parts of the body. The score is between 0-28. Higher scores indicate having more number of painful body regions.
Chair Test | 1 year
  In this test, which evaluates lower extremity muscle strength, participants sit and stand up as fast as possible for 30 seconds in a standard chair which is an average height of 44 cm and without back support and arm support. The number of repetitions which are completed were recorded
The Timed Up and Go Test | 1 year
  In this test, where functional mobility was evaluated, the evaluation was started while the participant was sitting in the chair. It recorded the time that a participant took to rise from a chair, walked three meters, turned around, walked back to the chair, and sat down
Single Leg Stance Test | 1 year
  This test evaluate participant's balance. The participant must stand unassisted on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground.
Tampa Kinesiophobia Scale | 1 year
  It is a 17-item scale that assesses fear of movement/ repeat injury. The range of total score are from 17 to 68. High score indicates that the person has high kinesiophobia
Fatigue Severity Scale | 1 year
  It was developed to evaluate the severity of fatigue in the last week. The range of total score are from 1 to 7. Higher scores indicate more severity of fatigue
Pittsburgh Sleep Quality Index | 1 year
  It was developed to identify good and poor sleep and to evaluate sleep quality. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5"or greater indicates a "poor" sleeper.
Cognitive Exercise Therapy Approach- Biopsychosocial Questionnaire | 1 year
  This scale, which was developed in Turkish and consists of 30 items, was used to evaluate the disease-related biopsychosocial process. The range of total score are from 0 to 120. Higher scores indicate bad biopsychosocial status of patients.
Short Form-36 | 1 year
  This scale is one of the most commonly used questionnaires to assess quality of life. "100 points" indicate good health status and "0 points" indicate poor health status.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Basakcı Calık, Assoc.Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University School of Physical Therapy and Rehabilitation, Denizli, Turkey (Türkiye)

REFERENCES:
- [Background] Ekici G, Unal E, Akbayrak T, Vardar-Yagli N, Yakut Y, Karabulut E. Effects of active/passive interventions on pain, anxiety, and quality of life in women with fibromyalgia: Randomized controlled pilot trial. Women Health. 2017 Jan;57(1):88-107. doi: 10.1080/03630242.2016.1153017. Epub 2016 Feb 16. PMID 26882533
- [Background] Altan L, Korkmaz N, Bingol U, Gunay B. Effect of pilates training on people with fibromyalgia syndrome: a pilot study. Arch Phys Med Rehabil. 2009 Dec;90(12):1983-8. doi: 10.1016/j.apmr.2009.06.021. PMID 19969158
- [Background] Silva HJA, Lins CAA, Nobre TTX, de Sousa VPS, Caldas RTJ, de Souza MC. Mat Pilates and aquatic aerobic exercises for women with fibromyalgia: a protocol for a randomised controlled blind study. BMJ Open. 2019 Feb 19;9(2):e022306. doi: 10.1136/bmjopen-2018-022306. PMID 30782866
- [Background] Franco KFM, Franco YRDS, Salvador EMES, do Nascimento BCB, Miyamoto GC, Cabral CMN. Effectiveness and cost-effectiveness of the modified Pilates method versus aerobic exercise in the treatment of patients with fibromyalgia: protocol for a randomized controlled trial. BMC Rheumatol. 2019 Jan 18;3:2. doi: 10.1186/s41927-018-0051-6. eCollection 2019. PMID 30886990
- [Derived] Caglayan BC, Basakci Calik B, Gur Kabul E, Karasu U. Investigation of effectiveness of reformer pilates in individuals with fibromyalgia: A randomized controlled trial. Reumatol Clin (Engl Ed). 2023 Jan;19(1):18-25. doi: 10.1016/j.reumae.2022.01.003. PMID 36603963